CLINICAL TRIAL: NCT01783054
Title: Pilot Study of Neoadjuvant Gemcitabine and Abraxane Chemotherapy Followed by Surgery for Patients With Localized, Resectable Adenocarcinoma of the Pancreas
Brief Title: Pilot, Neoadjuvant Gemcitabine and Abraxane Chemotherapy Followed by Surgery, Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study terminated due to low accrual
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101826
Record Dates: First submitted 2012-09-10; First posted 2013-02-04 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2015-10

CONDITIONS: Adenocarcinoma Pancreas
Keywords: NEOADJUVANT GEMCITABINE AND ABRAXANE CHEMOTHERAPY; SURGERY; RESECTABLE ADENOCARCINOMA OF THE PANCREAS
MeSH Terms: interventions — Surgical Procedures, Operative; Drug Therapy; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemotherapy, surgery, genetic expression (Experimental): All patients enrolled on study will start study treatment on a chemotherapy treatment regimen of Gemcitabine and abraxane. Treatment will be given on days 1, 8 and 15 of each cycle for 2 cycles over the course of 12 weeks.
  Patients will move on to surgery, 4-8 weeks after chemotherapy treatment. Patients must be recovered from any adverse effects of the chemotherapy before proceeding with surgery.
  As part of this study, tissue samples will be collect from each patient at the time of surgery for gene expression testing
  Interventions: Procedure: Surgery; Genetic: Genetic Expression; Drug: Chemotherapy

INTERVENTIONS:
Procedure: Surgery — Subjects will then receive surgery at MUSC within 4-8 weeks following completion of chemotherapy
Genetic: Genetic Expression — Subjects will have genetic expression testing done on their tissue samples.
Drug: Chemotherapy — Patients will receive gemcitabine at 1000 mg/m2 and abraxane at 125 mg/m2 intravenously on days 1, 8 and 15 of a 28 day cycle for 2 cycles
  Other Names: Gemcitabine; Abraxane

SUMMARY:
This study is for adult patients with adenocarcinoma of the pancreas. The purpose of this research study is to evaluate the safety and effectiveness of the drugs Gemcitabine and Abraxane in the treatment of adenocarcinoma of the pancreas before surgery. Subjects will have screening tests to determine if he or she is eligible to participate in this study.

DETAILED DESCRIPTION:
If subjects are eligible and wish to enroll in the study, they will begin chemotherapy treatment with Gemcitabine and Abraxane. After subjects have received treatment with these drugs, they will have surgery. Subjects will also have post treatment and follow up evaluations. Subjects may have 2 cycles of treatment and each cycle is 28 days. All subjects will be followed every 3 months for 3 years after their initial registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically or cytologically confirmed potentially resectable adenocarcinoma of the pancreas including tumors in the pancreatic head, uncinate process, neck, body and tail that are potentially resectable by pancreatico-duodenectomy (Kausch-Whipple procedure). Patients with islet cell or other neuroendocrine neoplasms are excluded.
* Definition of localized, potentially resectable disease:
* Staging by intravenous contrast-enhanced thin section helical abdominal computed tomography (2.5 mm cuts or less) or MRI (for patients with an IV contrast allergy) using pancreatic protocol. Endoscopic ultrasound is required for tissue acquisition and staging confirmation.
* No extension to superior mesenteric artery (SMA) and hepatic artery. Patent superior mesenteric vein/portal vein (SMV/PV) with < 180-degree abutment and no evidence of invasion.
* Clear fat plane between the SMA and celiac axis.
* No extension to celiac axis and hepatic artery.
* Patent superior mesenteric vein and portal vein.
* No evidence of distant disease.
* Male or non-pregnant and non-lactating female, and ≥ 18 years of age.
* If a female patient is of childbearing potential, she must have a negative serum pregnancy test documented within 72 hours of the first administration of study drug.
* If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator.
* Patient must not have received prior chemotherapy or radiation for pancreatic cancer.
* Patient has the acceptable blood counts as outlined in the protocol.
* Patient has an ECOG performance status PS 0-2.
* Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form prior to participation in any study-related activities.

Exclusion Criteria:

* Patient has borderline resectable, locally advanced unresectable or advanced metastatic disease. Patients with adenocarcinoma of the distal pancreatic body or tail are ineligible. Patients with endocrine tumors, lymphoma of the pancreas, or ampullary cancer are also ineligible.
* Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Patient has known infection with HIV.
* Patient has undergone major surgery, other than diagnostic surgery (i.e.surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
* Patient has a history of allergy or hypersensitivity to the study drugs.
* Patient has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive chemotherapy and/or radiation therapy.
* Patients requires chronic use of immunosuppressive agents (e.g. methotrexate, cyclosporine).
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for five years.
* Patients must not have clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) < 1 year before randomization.
* Patient is unwilling or unable to comply with study procedures.
* Patient is enrolled in any other therapeutic clinical protocol or investigational trial.
* Patients aged ≥ 80 are not excluded. However, candidates in this age group should be thoroughly evaluated before enrollment in the study, to ensure they are fit to receive chemotherapy, and to potentially undergo pancreaticoduodenectomy. In addition to meeting all of the baseline patient selection criteria, clinical judgment on their susceptibility to infection and expected stability of their performance status and suitability to receive intensive chemotherapy cycles, should be paid special attention to. Patients should not be enrolled in the study should there be any hesitation on any of these considerations. Baseline criteria for all patients enrolled on the study must be carefully evaluated and all criteria followed appropriately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kimchi, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy, Surgery: All subjects enrolled on study will start study treatment on a chemotherapy treatment regimen of Gemcitabine and abraxane. Gemcitabine and abraxane will be given on days 1, 8 and 15 of each cycle for 2 cycles over the course of 12 weeks, then surgery.
Period: Overall Study
Arm/Group | Chemotherapy, Surgery
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy, Surgery
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Estimate the rate of good histopathologic tumor response to neoadjuvant chemotherapy assessed in resection specimen. A good response is defined as a grade III or IV histopathologic appearance, equivalent to <10% viable tumor.
Time Frame: at time of surgery
Population: The study terminated early and the data for this outcome measure was not documented.
Arm/Group | Chemotherapy, Surgery
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With R0 Resection Status.
Description: R0 resection status is a macroscopic complete removal of tumor by non-contaminated operation, with neither macroscopic nor microscopic residual tumor.
Time Frame: at time of surgery
Population: Subjects who had surgical resection are included in the analysis for this endpoint.
Measure: Number; unit: participants
Arm/Group | Chemotherapy, Surgery
Number analyzed (Participants) | 2
participants | 2

3. Other Pre Specified Outcome: Circulating Tumor Cells (CTC)
Description: To evaluate and describe CTC number, CTC phenotype characteristics and effectiveness/rate of CTC culturing techniquen from patients with pancreatic adenocarcinoma. To determine and evaluate the correlation between expression of biomarkers in CTCs and expression of biomarkers in resected tissue specimen with the same cancer patient.
Time Frame: From enrollment to surgery
Population: This outcome measure was added as part of an amendment. No subjects were enrolled after this amendment was instituted, so no outcomes measures were collected.
Arm/Group | Chemotherapy, Surgery
Number analyzed (Participants) | 0

4. Secondary Outcome: Estimate Median Time to Recurrence.
Description: Time to recurrence is defined as the time from surgical resection to disease recurrence or death from any cause. Patients who have not recurred at the end of follow up will have their recurrence time censored at the last date of contact.
Time Frame: 2 years
Population: Only subjects who had surgical resection are included in the analysis for this endpoint. At the time of these results, one subject expired due to disease progression. The other subject was still alive at the time of termination, so is not included in the outcome measure data below.
Measure: Number; unit: days
Arm/Group | Chemotherapy, Surgery
Number analyzed (Participants) | 1
days | 329

5. Secondary Outcome: Estimate Median Overall Survival
Description: Overall survival is defined as the time from enrollment to death from any cause. Patients still alive at the end of follow up will have their survival time censored at the last date of contact.
Time Frame: 2 years
Population: as for outcome 4
Measure: Number; unit: days
Arm/Group | Chemotherapy, Surgery
Number analyzed (Participants) | 1
days | 465

6. Secondary Outcome: Number of Adverse Events Reported in Subjects Enrolled.
Description: Assess the safety profile of this neoadjuvant regimen in patients with localized pancreatic adenocarcinoma. All toxicities will be reported by type and grade and tabulated. All adverse events will be reported via case report forms. The intensity of any adverse event should be reported according to the NCI Common Terminology Criteria for Adverse Events v4.0.
Time Frame: First study drug administration until end of study
Population: All subjects who were administered study intervention and had documented adverse events were analyzed. The number below represents the number of adverse events, including serious adverse events, reported on by enrolled subjects. A complete list of the adverse events reported are in the adverse events tables of these results.
Measure: Number; unit: adverse events
Arm/Group | Chemotherapy, Surgery
Number analyzed (Participants) | 2
adverse events | 60

ADVERSE EVENTS:
Arm/Group | Chemotherapy, Surgery
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy, Surgery (N=2)
cholangitis (Hepatobiliary disorders) | 1 (1)
biliary stent drainage (Hepatobiliary disorders) | 1 (1)
renal insuffiency (Renal and urinary disorders) | 1 (1)
fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy, Surgery (N=2)
anemia (Blood and lymphatic system disorders) | 2 (2)
hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 1 (1)
aortic valve disease (Cardiac disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1)
flatulence (Gastrointestinal disorders) | 1 (1)
edema limb (General disorders) | 2 (2)
flu like symptoms (General disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
pain (General disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 1 (1)
biliary anastomic leak (Injury, poisoning and procedural complications) | 1 (1)
wound complication (Injury, poisoning and procedural complications) | 1 (1)
ALT increased (Investigations) | 2 (2)
AST increased (Investigations) | 2 (2)
creatinine increased (Investigations) | 2 (2)
alkaline phosphatase increased (Investigations) | 1 (1)
blood bilirubin increased (Investigations) | 1 (1)
lymphocyte count decreased (Investigations) | 1 (1)
neutrophil count decreased (Investigations) | 1 (1)
platelet count decreased (Investigations) | 1 (1)
urine output decreased (Investigations) | 1 (1)
weight loss (Investigations) | 1 (1)
white blood cell decreased (Investigations) | 1 (1)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
hypokalemia (Investigations) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
neck pain (Metabolism and nutrition disorders) | 1 (1)
agitation (Metabolism and nutrition disorders) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1)
urine discoloration (Renal and urinary disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes